CLINICAL TRIAL: NCT03855579
Title: Levosimendan Versus Milrinone to Support Hemodynamics During Off Pump Coronary Artery Bypass Grafting Surgery in Patients With Poor Ejection Fraction
Brief Title: Levosimendan Versus Milrinone in Off Pump CABG Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hany Mostafa Esmaeil Osman, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Levosimendan, Milrinone, CABG
Record Dates: First submitted 2019-02-24; First posted 2019-02-27 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Hemodynamics
Keywords: Levosimendan; Milrinone; Off-pump; Coronary
MeSH Terms: interventions — Simendan; Milrinone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levosimendan (Experimental): Intraoperative infusion of Levosimendan
  Interventions: Drug: Levosimendan
- Milrinone (Active Comparator): Intraoperative infusion of Milrinone
  Interventions: Drug: Milrinone

INTERVENTIONS:
Drug: Levosimendan — Intraoperative infusion of Levosimendan
  Arms: Levosimendan
Drug: Milrinone — Intraoperative infusion of Milrinone
  Arms: Milrinone

SUMMARY:
To compare the efficacy of Levosimendan versus Milrinone in supporting hemodynamics during off-pump coronary artery bypass grafting surgery in patients with low ejection fraction.

DETAILED DESCRIPTION:
The major challenge during off-pump coronary artery bypass graft surgery is to maintain optimum hemodynamics by optimizing the intravascular volume and by using some inotropes. However, conventional inotropes such as beta-agonists are associated with tachycardia and arrhythmia which increase myocardial oxygen demand.

Levosimendan is an inodilator which exerts its positive inotropic effect by enhancing the sensitivity of troponin C to calcium without increasing intracellular calcium concentration. Levosimendan also decreases the systemic vascular resistance, so, it increases the cardiac output without increasing myocardial oxygen consumption.

This study aims to compare the efficacy of Levosimendan versus Milrinone in supporting hemodynamics during off-pump coronary artery bypass grafting surgery in patients with low ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Elective off-pump coronary artery bypass grafting surgery.
* ejection fraction < 50%

Exclusion Criteria:

* Patients with severe renal impairment or renal failure.
* Patients on mechanical support (intra-aortic balloon pump)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-09-10 (Estimated); Study Completion 2019-09-10 (Estimated)

PRIMARY OUTCOMES:
Mean blood pressure | Intraoperative
Consumption of other inotropes | Intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided